CLINICAL TRIAL: NCT04757818
Title: Double-blind, Randomized, Parallel, Placebo-controlled Clinical Study to Evaluate the Viral Load of SARS-CoV-2 in the Oral Cavity of SARS-CoV-2 Positive Subjects After the Use of a Mouthwash Containing Cetylpyridinium Chloride 0,07%
Brief Title: Double-blind, Randomized, Parallel, Placebo-controlled Clinical Study to Evaluate the Viral Load of SARS-CoV-2 (COVID-19) in the Oral Cavity of SARS-CoV-2 Positive Subjects After the Use of a Mouthwash Containing Cetylpyridinium Chloride 0,07%.
Acronym: CPC COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentaid SL (Industry)
Collaborators: IrsiCaixa (Other); Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CPC COVID
Record Dates: First submitted 2021-02-16; First posted 2021-02-17 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; Cetylpyridinium chloride; COVID19; Mouthwash; Saliva sample; RT-qPCR
MeSH Terms: conditions — COVID-19 | interventions — Cetylpyridinium; cytidylyl-(3'-5')-cytidine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, parallel, placebo-controlled clinical study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.07% cetylpyridinium chloride (CPC) in mouthwash (Experimental): Single dose. A mouthwash and gargles with 15 ml of product for 1 minute.
  Interventions: Other: 0.07% cetylpyridinium chloride (CPC) in mouthwash
- Distilled water with the same colorant as the experimental product (Placebo Comparator): Single dose. A mouthwash and gargles with 15 ml of product for 1 minute.
  Interventions: Other: Distilled water with the same colorant as the experimental product

INTERVENTIONS:
Other: 0.07% cetylpyridinium chloride (CPC) in mouthwash — A mouthwash and gargles with 15 ml of 0.07% cetylpyridinium chloride (CPC) in mouthwash for 1 minute.
  Arms: 0.07% cetylpyridinium chloride (CPC) in mouthwash
Other: Distilled water with the same colorant as the experimental product — A mouthwash and gargles with 15 ml of distilled water for 1 minute
  Arms: Distilled water with the same colorant as the experimental product

SUMMARY:
Double-blind, parallel, randomized, placebo-controlled clinical study. Subjects with confirmed SARS-CoV-2 infection by PCR or antigen rapid test, asymptomatic or with mild COVID-19 symptoms will be included. Subjects who agree to participate and who are eligible will be randomized to perform a mouth rinse and gargle with a 0.07% CPC mouthwash (experimental) or with a substance of the same color (placebo). Saliva samples will be collected at baseline (i.e., before wash) and 1 hour and 3 hours after wash. Saliva samples will be transferred to a central laboratory for SARS-CoV-2 viral load determination, nucleocapsid protein levels determination, rapid antigen testing, viral infectivity analysis and storage.

DETAILED DESCRIPTION:
Study procedures will be as follows:

The study procedures will take place in 1 day (total interval of 3 hours from the baseline sample collection to the last sample collection).

The study samples will be saliva samples (1-1.5 ml) collected at baseline and 1 and 3 hours after the intervention. The intervention will be the use of a mouthwash (washes and gargles) for one minute with 15 ml of either CPC Protect® (CPC group) or colored distilled water (control group).

Candidates with a positive result of PCR or antigen rapid test for SARS-CoV-2 will be identified by study nurses, certified nursing assistants, and dentists at primary health care centers of the Metro Nord health administrative region of Catalonia. The investigator will obtain the candidates' informed consent and will verify that the subject meets all the inclusion criteria and none of the exclusion criteria. The researcher will assign a correlative kit number (randomization) and instruct the subject in the procedure of self-collection of a saliva sample.

Baseline: The subject will self-collect the baseline saliva sample in front of the investigator, who will be able to correct the errors observed in the procedure.

Hour 0: After the obtention of the baseline saliva sample, the subject will rinse and gargle with 15 mL of mouthwash (experimental or placebo) for 1 minute (30 seconds of rinsing and 30 seconds of gargling).

The researcher will indicate to the subject the hours in which the second and third saliva samples should be taken. The subject must avoid brushing their teeth, eating and drinking, except water, until the rest of the saliva samples are collected and may return home.

Hour 1: One hour after mouthwash use, the subject will self-collect the second saliva sample (1-hour sample).

Hour 3: Three hours after mouthwash use, the subject will self-collect the third saliva sample (3-hour sample).

The investigator will contact the subject to confirm the correct collection of saliva samples (1 hour and 3 hours) at the indicated times and will record it in the study application.

Saliva samples will be collected at the center and/or at the subjects' residence and will be transferred to the Clinical Laboratory Metropolitana Nord in Hospital Universitari Germans Trias i Pujol (HUGTiP) for the viral load analysis by RT-PCR. The remaining saliva volume will be transferred to IrsiCaixa's Laboratory (located in the HUGTiP) for the ELISA analysis and the rest of the analysis, and for storage in those cases where the subject's IC is available for it.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or greater than 18 years
2. 2. Confirmation of SARS-CoV-2 infection, determined by PCR or validated rapid antigen test1 from a nasopharyngeal smear performed in ≤3 days.
3. Without symptoms of COVID-19 or with symptoms with ≤3 days of evolution
4. Cognitive and motor ability to perform mouthwashes and gargles
5. Willingness to comply with the requirements of the protocol
6. Understanding of the information provided in relation to the objectives and procedures
7. Provide your consent freely to participate in the study.

Exclusion Criteria:

1. Use of mouthwashes, in the last 24 hours
2. Use of VITIS pastes and / or PERIO AID gel, in the last 24 hours
3. Four or more days of symptoms compatible with COVID-19.
4. Recent medical diagnosis (≤ 1 month) of pneumonia
5. Cognitive impairment or other reason that, in the investigator's discretion, contraindicates participation in the study
6. Hyposialia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 viral load in saliva samples measured by RT-qPCR | 1 hour and 3 hours after intervention
  To determine the efficacy of a 0.07% CPC mouthwash in reducing the viral load of SARS-CoV-2 in saliva samples, measured by RT-qPCR, in subjects with confirmed SARS-CoV-2 infection
Nucleocapsid protein levels in saliva samples measured by ELISA | 1 hour and 3 hours after intervention
  To determine the efficacy of a 0.07% CPC mouthwash in increasing the nucleocapsid protein levels in saliva samples, measured by high-sensitivity quantitative ELISA (ImmunoDiagnostics), in subjects with confirmed SARS-CoV-2 infection

SECONDARY OUTCOMES:
SARS-CoV-2 viral load in saliva samples determined by RT-qPCR | 1 hour after intervention
  To determine the reduction of SARS-CoV-2 viral load by RT-qPCR in saliva samples
SARS-CoV-2 viral load in saliva samples determined by RT-qPCR | 3 hours after intervention
  To determine the reduction of SARS-CoV-2 viral load by RT-qPCR in saliva samples
Sensitivity and specificity of different rapid SARS-CoV-2 antigen tests compared to RT-qPCR in saliva samples | 1 hour and 3 hours after intervention
  To compare the sensitivity and specificity of rapid SARS-CoV-2 antigen tests compared to RT-qPCR in saliva samples
Intraindividual difference in SARS-CoV-2 infectivity in vitro before and after treatment with a 0.07% CPC or placebo | Baseline, 1 hour and 3 hours after intervention
  To determine the intraindividual difference in SARS-CoV-2 infectivity in vitro before and after treatment with a 0.07% CPC or placebo

CONTACTS AND LOCATIONS:
Locations (19):
- Spain (19):
  - CAP Gorg, Badalona, Barcelona
  - CAP Gran Sol, Badalona, Barcelona
  - CAP St Roc, Badalona, Barcelona
  - CAP Barri Llatí, Santa Coloma de Gramenet, Barcelona
  - CAP Fondo, Santa Coloma de Gramenet, Barcelona
  - CAP Santa Rosa, Santa Coloma de Gramenet, Barcelona
  - CAP Singuerlin, Santa Coloma de Gramenet, Barcelona
  - CAP Dr Robert, Badalona
  - CAP Les Franqueses del Vallès, Bellavista
  - CAP Canovelles/Granollers Oest, Canovelles
  - CAP Granollers Centre, Granollers
  - ABS Gatassa, Mataró
  - EAP Mollet Est, Mollet del Vallès
  - CAP Montornés/Montmeló, Montornés Del Vallès
  - CAP Palau, Palau-solità i Plegamans
  - EAP Parets del Vallès, Parets del Vallès
  - CAP Sant Celoni, Sant Celoni
  - CAP Santa Perpètua, Santa Perpètua de Mogoda
  - EAP Vilassar de Mar, Vilassar de Mar